CLINICAL TRIAL: NCT00302978
Title: The Effects of in Vivo Exposure Therapy on the Neural Correlates of Height Phobia: a Functional Magnetic Resonance Imaging Study Using a Fear Provocation Paradigm.
Brief Title: Changes in Brain Activity (Functional MRI Study) Before and After Behavioral Therapy of Height Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5215
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2007-04

CONDITIONS: Height Phobia; Fear of Heights
Keywords: Height phobia; fear of heights; specific phobia
MeSH Terms: conditions — Acrophobia; Phobia, Specific | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior therapy

SUMMARY:
We are interested in investigating the functional brain abnormalities of height phobia. Subjects will be have a functional MRI scan before and after a course of treatment with behavioral therapy.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of in vivo exposure therapy on the functional brain activity of subjects with height phobia using a fear provocation paradigm. We expect differential activation of the fear circuitry in height phobics compared to non-phobic controls, and that successful behavioral therapy will normalize the heightened fear response in height phobia.

ELIGIBILITY:
Inclusion Criteria:

* Specific phobia of Heights

Exclusion Criteria:

* History of medical problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-03; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
CGI

SECONDARY OUTCOMES:
acrophobia questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yujuan Choy, M.D., Principal Investigator — New York State Psychiatric Institute, Columbia University